CLINICAL TRIAL: NCT01310348
Title: Effect of Bone Mineral Density on Vibration-Induced Muscle Strength Gain at The Lower Limbs
Brief Title: Effect of Bone on Vibration-Induced Muscle Strength Gain
Acronym: EBVIMSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Karacan, Chief of Physical Med & Rehab Clinic, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BEAH FTR-2
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Bone Mass; Effects of Vibration
Keywords: Bone; Muscle strength; whole-body vibration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very low magnitude vibration (Placebo Comparator): Very low magnitude vibration
  Interventions: Device: WBV (Sham stimulation)
- Training (Experimental): The whole-body vibration (WBV) training
  Interventions: Device: whole-body vibration (WBV)

INTERVENTIONS:
Device: whole-body vibration (WBV) — The whole-body vibration (WBV) training group will be trained on a WBV platform (Power Plate) 5 times a week for 4 weeks period. Training volume and training intensity will be low at the beginning but progressed slowly according to the overload principle. The training volume will be increased systematically over the 4-week training period. The training intensity will be increased by increasing the amplitude (2-4 mm) and the frequency (40 Hz) of the vibration.
  Other Names: Cyclic mechanical loading
  Arms: Training
Device: WBV (Sham stimulation) — Sham stimulus will be performed by WBV platform 5 times a week for a 4 weeks period.
  Arms: Very low magnitude vibration

SUMMARY:
The aim of this study is to investigate whether there is a relation between bone mineral density of lower limbs exposed to vibration and the muscle strength gain in the knee extensors and flexors, and a relation serum sclerostin level and the muscle strength gain in the knee extensors and flexors in healthy young adult women.

Forty healthy young adult women are planned to include in this study. The participants meeting the criteria were randomized into two groups: the training group (20 cases) and the Control group (20 cases).

The whole-body vibration (WBV) training group will be trained on a WBV platform (Power Plate) 5 times a week for 4 weeks period. Participants will be asked to stand upright on WBV platform. Training volume and training intensity will be low at the beginning but progressed slowly according to the overload principle. The training volume will be increased systematically over the 4-week training period. The training intensity will be increased by increasing the amplitude (2-4 mm) and the frequency (40 Hz) of the vibration. The subjects will be asked to report negative side effects or adverse reactions in their training diary. In the Control group, sham stimulus will be performed by WBV platform 5 times a week for a 4 weeks period.

Plasma sclerostin level and, the right and left knee flexor and extensor muscles strength will be measured before and after training period. Isokinetic torque will be measured with the Biodex (Biodex System 3 PRO Multijoint System Biodex Medical Inc. Shirley/NY USA)extremity-testing system. The right and left lower limbs bone mineral density (BMD) and muscle strength will be measured before training period. The BMD will be evaluated by bone densitometer (Norland XR-46 DXA, USA). Sclerostin levels will be measured by human sclerostin ELISA kit.

The rest muscle electrical activity of right and left knee flexor and extensor muscles will be evaluated at pre-vibration, post- vibration and, during vibration. The rest muscle electrical activity will be measured by Powerlab (data acquisition system, ADInstruments, Australia) device.

DETAILED DESCRIPTION:
Vibration has a strong osteogenic effect. Vibration-induced bone formation is neuronally regulated. Vibration can also effectively enhance muscle strength and power. Previous studies have shown that vibration increases muscle electromyographic (EMG) activity. Attempts to explain vibration-induced increases in EMG activity were based on the tonic vibration reflex. Tonic vibration reflex activates the muscle spindles, thereby enhancing the excitatory drive reflex of the alpha motoneurons. On the contrary, it was shown that the vibration treatment did not enhance the muscle spindle sensitivity and led to presynaptic inhibition of muscle spindle group Ia afferents. As an alternative to tonic vibration reflex, the recently described bone myoregulation reflex has been suggested to potentially explain the increased muscle strength and electrical activity induced by vibration. Based on the bone myoregulation reflex, bone is sensitive to mechanical stimuli and can send mechanical input signals to central nervous system and so can neuronally regulate the muscle activity.

The cyclic mechanical loading to the bone stimulates the osteocytes. According to bone myoregulation reflex, the more the osteocytes are stimulated by the cyclic mechanical loading, the increase occurring in the muscle strength and activity may be more. The rate of osteocytes stimulated by vibration may be determined with serum sclerostin level. Sclerostin, the protein product of the SOST gene, is an osteocyte-specific cysteine knot-secreted glycoprotein that is a potent inhibitor of bone formation. Sost/sclerostin levels have been reported to be reduced by mechanical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women,
* Women with ages varying between 20 and 40 years
* Right-handed women

Exclusion Criteria:

* Bone, muscle/tendon, joint, vascular, dermatologic diseases in lower extremities and spine
* Medication that could affect the musculoskeletal system
* Postural abnormalities (scoliosis, kyphosis, etc)
* Systemic diseases

  * Hypertension ( Diastolic > 85 mmHg, Systolic>135 mmHg)
  * Heart Diseases (coronary heart disease, conduction or rhythmic problems, pacemaker etc.)
  * Abdominal disease (Gallstone etc)
  * Urinary disease (kidneystone etc)
  * Gynecological disease (menstrual irregularities, etc)
  * Infectious disease
  * Endocrine diseases such as diabetes mellitus or other disease
* Neurologic disorders (central or peripheral)
* Pregnancy or lactation
* Obesity (BMI >30 kg/m2 or body weight > 80 kg )
* Vertigo
* Cognitive dysfunction
* Professional/regular sports activity and heavy worker

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Vibration-induced muscle strength gain | 6 months
  Effects of bone mineral density on vibration-induced muscle strength gain

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Cidem M, Karacan I, Diracoglu D, Yildiz A, Kucuk SH, Uludag M, Gun K, Ozkaya M, Karamehmetoglu SS. A Randomized Trial on the Effect of Bone Tissue on Vibration-induced Muscle Strength Gain and Vibration-induced Reflex Muscle Activity. Balkan Med J. 2014 Mar;31(1):11-22. doi: 10.5152/balkanmedj.2013.9482. Epub 2014 Mar 1. PMID 25207162